CLINICAL TRIAL: NCT01095276
Title: Inhaled Dnase (Pulmozyme®) as a Non-Invasive Treatment of Atelectasis in Mechanically Ventilated Patients
Brief Title: Impact of Nebulized Dornase Alpha on Mechanically Ventilated Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Responsible Party: Jessica Nutik Zitter, MD, MPH, University of Medicine and Dentistry of New Jersey
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0120030304
Record Dates: First submitted 2009-07-28; First posted 2010-03-30 (Estimated); Last update posted 2010-03-30 (Estimated); Status verified 2010-03

CONDITIONS: Atelectasis; Ventilation, Mechanical
Keywords: Mechanical Ventilation; Extubation; dornase alpha; oxygenation; chest x ray
MeSH Terms: conditions — Pulmonary Atelectasis; Respiratory Aspiration | interventions — dornase alfa; Deoxyribonucleases; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nebulized saline (Placebo Comparator): patients on mechanical ventilation who were randomized to receive a placebo comparator (vehicle solution for dornase alpha)
  Interventions: Drug: Saline
- dornase alpha (Active Comparator): patients on mechanical ventilation who were randomly assigned to receive dornase alpha by in-line nebulization
  Interventions: Drug: Pulmozyme (nebulized dornase alpha)

INTERVENTIONS:
Drug: Pulmozyme (nebulized dornase alpha) — nebulized dornase alpha: 2.5 mg by in-line nebulizer BID
  Other Names: Pulmozyme; DNase
  Arms: dornase alpha
Drug: Saline — Saline packaged identically to the dornase alpha intervention unit doses and coded for blinding by the company providing the intervention drug (dornase alpha).
  Arms: Nebulized saline

SUMMARY:
The investigators hypothesized that dornase alpha, administered twice a day (BID) by in-line nebulizer, would improve oxygenation, compliance, and time to extubation in adult patients receiving mechanical ventilation.

DETAILED DESCRIPTION:
Background: Lobar or segmental collapse of the lung in mechanically ventilated patients is a relatively common occurrence in the Intensive Care Unit. Available treatments are either labor or time intensive and not highly effective.

Methods: We conducted a randomized, placebo-controlled, double-blind pilot study to determine whether nebulized recombinant human dornase alpha (Pulmozyme, Genentech) improves radiologic and clinical outcomes in ventilated patients with lobar atelectasis. Outcomes of interest were chest radiograph score, oxygenation, lung compliance, and rate of extubation over the first 5 days. The groups consisted of 14 intervention patients and 16 control patients. They were similar with respect to basic demographics, age, gender, and use of therapeutic modalities relating to lung function. Baseline average chest x-ray scores, Pa02/FI02 ratios, and static compliance were not significantly different. Analysis was limited to the first 5 days.

Results: There was a significant improvement in oxygenation for the intervention group at day 5 (p=0.03). There were no significant differences in chest radiograph score, compliance, or rate of extubation. Two patients died in the intervention group, whereas none died in the control group (NS).

Conclusions: These pilot data suggest that inhaled dornase alpha appears to be safe and is associated with improved oxygenation 5 days after initiation of therapy in mechanically ventilated patients compared to placebo. Larger studies are needed to confirm these findings and determine if this intervention decreases ICU morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* current ventilator use
* onset of lobar or whole lung collapse over the previous 12 hours
* age greater than 18

Exclusion Criteria:

* quadriplegia or debilitating neuromuscular condition
* chronic ventilator dependence
* pneumothorax
* frank hemoptysis
* elevated intracranial pressure
* intracranial bleed
* pregnancy or active nursing
* concurrent use of other investigational drugs
* history of allergy to Pulmozyme®, Chinese Hamster Ovary-derived biologics, or any of the components of the active or placebo formulations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-11; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Total Chest X Ray Score | Days 0-30

SECONDARY OUTCOMES:
Oxygenation (Pa02/FI02) | Days 0-30
Static Lung Compliance | Days 0-30
Time to Extubation | Days 0-30

CONTACTS AND LOCATIONS:
Overall Officials: Jessica N Zitter, MD, MPH, Principal Investigator — UMDNJ, Department of Medicine
Locations (1):
- University of Medicine and Dentistry of New Jersey, Newark, New Jersey, United States